Intramuscular Heating Rates of a Chattanooga Intelect XT Therapeutic Ultrasound with a 3 MHz frequency and 1.0 W/cm² Intensity at Three Depths up to 2.5 cm.

## Statistical Analysis Plan:

Twenty-five subjects will be recruited from the Institution's student population using the University email Listserv. Descriptive statistics will be utilized to determine the rate of increase for each depth. A 3 x 4 repeated measures ANOVA will be used to determine differences in temperature increases at 3 depths (1.0, 1.75 and 2.5 cm) at 4 different time points (baseline, 5,10,15 minutes). The level of significance will be set at  $p \le .05$